CLINICAL TRIAL: NCT01615978
Title: A Randomised, Double-blind Within Dose Group, Single-centre, Placebo-controlled, Parallel 2-different Dose Group, 14-day Multiple s.c. Doses Study to Assess the Safety, Pharmacokinetics and Pharmacodynamics of Liraglutide (NNC 90-1170) in Subjects With Type 2 Diabetes
Brief Title: Safety and Tolerability of Liraglutide in Japanese Subjects With Type 2 Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NN2211-1591
Record Dates: First submitted 2012-06-07; First posted 2012-06-11 (Estimated); Last update posted 2017-01-25 (Estimated); Status verified 2017-01

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — Liraglutide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fixed dose: 5 mcg/kg (Experimental)
  Interventions: Drug: liraglutide; Drug: placebo
- Escalated dose: 10 mcg/kg (Experimental)
  Interventions: Drug: liraglutide; Drug: placebo

INTERVENTIONS:
Drug: liraglutide — 5 mcg/kg daily for 14 days. Injected subcutaneously once daily
  Arms: Fixed dose: 5 mcg/kg
Drug: liraglutide — Initial dose of 5 mcg/kg for 7 days followed by 10 mcg/kg for 7 days. Injected subcutaneously once daily
  Arms: Escalated dose: 10 mcg/kg
Drug: placebo — Liraglutide placebo administered to subjects randomised at each dose level in the ratio of 3:1

SUMMARY:
This trial is conducted in Japan. The aim of this trial is to assess the safety after multiple s.c. (subcutaneously) doses of liraglutide in Japanese subjects with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes
* Duration of diabetes for more than 12 weeks
* Subjects currently on diet therapy (OHA-naïve) or treated with OHA (oral hypoglycaemic agent)
* monotherapy for more than 12 weeks
* HbA1c (Glycated haemoglobin A1c) between 6.0-9.0 %, both inclusive
* Body Mass Index (BMI): 18.5-30.0 kg/m^2

Exclusion Criteria:

* Recurrent severe hypoglycaemia
* Proliferative retinopathy or maculopathy requiring acute treatment
* Impaired hepatic function
* Impaired renal function
* Cardiac problems
* Uncontrolled treated/untreated hypertension
* Current treatment with insulin preparations or TZDs (thiazolidinediones)
* Current treatment or expected at the screening to start treatment with systemic corticosteroids

Ages: 20 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2003-12; Primary Completion 2004-03 (Actual); Study Completion 2004-03 (Actual)

PRIMARY OUTCOMES:
24-hour profiles of serum calcitonin
24-hour profiles of Ca2+ (ionised calcium)
24-hour profiles of PTH (Parathyroid Hormone)
Adverse events

SECONDARY OUTCOMES:
Area under the plasma liraglutide curve
Cmax, maximum plasma liraglutide concentration
tmax, time to reach Cmax
Terminal phase elimination rate-constant
t½, terminal elimination half life
24-hour profiles of serum insulin
24-hour profiles of plasma glucose

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Tokyo, Japan

REFERENCES:
- [Result] Kageyama S, Hirao K, Shimizu A, Matsumura Y, Zdravkovic M, Rasmussen MF, Irie S. Tolerability, pharmacokinetics, and pharmacodynamics of liraglutide, long-acting human GLP-1 analogue - Phase 1 studies in Japanese healthy subjects with type 2 diabetes. Endocrinology and Diabetology 2007; 24 (6): 95-104
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com